CLINICAL TRIAL: NCT05206448
Title: Randomized Controlled Trial of Combined Letrozole and Clomid (CLC II) Versus Letrozole Alone for Women With Anovulation
Acronym: CLC II
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rachel Mejia (Other)
Collaborators: Society for Reproductive Investigation (Unknown); American Society for Reproductive Medicine (Unknown); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor-Investigator, Rachel Mejia, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201906826
Record Dates: First submitted 2021-12-28; First posted 2022-01-25 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Polycystic Ovary Syndrome; PCOS; Infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Letrozole; Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole (Active Comparator): Letrozole 2.5 mg orally for 5 days on cycle days 3-7 in first study treatment cycle. Participants who ovulate and do not become pregnant will repeat the same treatment protocol for their next study cycle. Participants who do not ovulate will repeat the protocol with Letrozole dose increase of 2.5 mg daily in the next treatment cycle, to a maximum dose of 7.5 mg in the 3rd cycle.
  Interventions: Drug: Letrozole
- Letrozole + Clomiphene Citrate (Experimental): Letrozole 2.5 mg orally for 5 days on cycle days 3-7 AND Clomiphene Citrate 50 mg orally for 5 days on cycle days 3-7. Participants who ovulate and do not become pregnant will repeat the same treatment protocol for their next study cycle. Participants who do not ovulate will repeat the protocol with Letrozole dose increase of 2.5mg daily in the next treatment cycle to a maximum dose of 7.5 mg in the 3rd cycle, while maintaining the same dose of Clomiphene Citrate.
  Interventions: Drug: Letrozole; Drug: Clomiphene Citrate

INTERVENTIONS:
Drug: Letrozole — Letrozole tablet
  Other Names: femara
Drug: Clomiphene Citrate — Clomiphene Citrate tablet
  Other Names: Clomid; Clomiphene
  Arms: Letrozole + Clomiphene Citrate

SUMMARY:
This study evaluates the addition of clomiphene citrate (CC) to letrozole for the treatment of infertility in women with polycystic ovary syndrome across a course of two treatment cycles with stair step dosing of letrozole similar to standard of care. Half of the participants will receive letrozole and CC in combination, while the other half will receive letrozole alone.

DETAILED DESCRIPTION:
Letrozole and Clomid are both used for ovulation induction, but they have different mechanisms of action. In a pilot study we found that the combination of letrozole 2.5 mg and CC 50 mg nearly doubled the ovulation rate as compared to use of letrozole monotherapy (77% vs. 43%, P=0.007; rate ratio for ovulation (95% CI) 1.80 (1.18 to 2.75), with similar endometrial thickness and number of follicles across treatment arms among those who ovulated. Additional data is needed to evaluate escalating dosages, multiple cycles, live birth and multiple gestation with this novel treatment combination.

This is a randomized controlled trial of letrozole versus letrozole and clomiphene citrate (CC) for up to three menstrual cycles. Women will be randomized in a 1:1 ratio to receive letrozole 2.5 mg or combination of letrozole 2.5 mg and clomiphene 50 mg for 5 days on days 3-7 of menstrual cycle. The women and their partners will be instructed to have regular intercourse with the intent to conceive during the cycle. Patients will have an transvaginal ultrasound in the mid-luteal phase of cycle to assess corpora lutea number and endometrial thickness. Patients will have mid- luteal phase progesterone level drawn to evaluate ovulation. Patients in both study arms who do not ovulate will have their Letrozole dose increased by 2.5 mg in the next study cycle to a max of 7.5 mg. Patients in the combination arm who do not ovulate will only have their Letrozole dose increased and will continue to receive the same dose of clomiphene across the three study treatment cycles. Side effect profile will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to comply with all study procedures and be available for the duration of the study
2. Diagnosis of infertility: Inability of couple to achieve successful pregnancy after 12 months of regular time unprotected intercourse in women less than 35 years of age; and after 6 months of regular intercourse without use of contraception in women 35 years and older. Women that have anovulation or oligomenorrhea are also considered to meet diagnosis of infertility, without meeting the time constraints described above.
3. Diagnosis of polycystic ovary syndrome based on Revised Rotterdam criteria.
4. Ability to have regular intercourse during the ovulation induction phase of the study.
5. Partner with a normal sperm concentration of 15 million/mL and with normal motility of >40% according to World Health Organization cutoff points or greater than 10 million total motile sperm count OR has fathered a pregnancy in the past.

Exclusion Criteria:

1. Current pregnancy
2. Current use of hormonal contraception; use of any type of combined contraceptive or oral progestins within the past month; or use of hormonal implants or depo progestins within the past 3 months
3. Other known cause of infertility: endometriosis, tubal factor, uterine abnormalities
4. Uncorrected thyroid disease
5. Untreated hyperprolactinemia
6. Medical conditions in which avoiding pregnancy is recommended until under improved control: poorly controlled Type 1 or Type 2 diabetes, poorly controlled hypertension
7. Contraindications to clomiphene citrate: hypersensitivity to clomiphene citrate or any of its components, history of liver disease or known liver disease, unknown cause of abnormal uterine bleeding, or intracranial lesion
8. Contraindications to letrozole: hypersensitivity to letrozole or any of its components
9. Use of medications known to affect reproductive function or metabolism or that are an absolute contraindication during pregnancy within the past month
10. If patients are suspected based on clinical findings for other etiologies that mimic PCOS, work up must be completed to exclude other etiologies prior to enrollment (i.e. Cushing's syndrome, androgen-secreting tumor)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Mejia, DO, Principal Investigator — University of Iowa Hospitals & Clinics
Locations (4):
- United States (4):
  - University of Iowa Hospitals & Clinics - Davenport Clinic, Davenport, Iowa
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Iowa Hospitals & Clinics- West Des Moines Clinic, West Des Moines, Iowa
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate
Started | 98 | 92
Completed 1st Treatment Cycle | 98 | 92
Ongoing Pregnancy Resulting From Cycle 1 (Participants with ongoing pregnancy resulting from cycle 1 did not complete cycle 2 or 3 per protocol and were considered as completing study participation.) | 4 | 15
Completed 2nd Treatment Cycle (Participants with ongoing pregnancy resulting from cycle 1 did not complete additional treatment cycles.) | 93 | 75
Ongoing Pregnancy Resulting From Cycle 2 (Participants with an ongoing pregnancy from cycle 2 did not complete cycle 3 per protocol and were considered as completing study participation.) | 10 | 8
Completed 3rd Treatment Cycle (Participants with ongoing pregnancy resulting from cycle 1 or 2 did not complete additional treatment cycle) | 78 | 65
Completed | 92 (Sum of those who completed 3 treatment cycles, those who had an ongoing pregnancy from treatment cycle 1 and those who had an ongoing pregnancy in treatment cycle 2.) | 88 (Sum of those who completed 3 treatment cycles, those who had an ongoing pregnancy from treatment cycle 1 and those who had an ongoing pregnancy in treatment cycle 2.)
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — found ineligible after randomization | 1 | 1
Not completed — unable to complete study due to personal constraints | 1 | 0
Not completed — Became pregnant during gap in treatment after pregnancy loss | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate | Total
Number analyzed (Participants) | 98 | 92 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (4.25) | 29.9 (4.31) | 30.2 (4.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 92 | 190
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-hispanic | 79 | 79 | 158
  Black non-hispanic | 3 | 1 | 4
  Asian | 4 | 2 | 6
  Hispanic | 10 | 7 | 17
  Multiple | 1 | 2 | 3
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 98 | 92 | 190
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.24 (7.97) | 36.78 (7.91) | 36.50 (7.92)

OUTCOME MEASURES:

1. Primary Outcome: Ovulation
Description: Number of Participants with Mid-luteal serum progesterone level >=3 ng/ml Number of cycles with Mid-luteal serum progesterone level >=3 ng/ml
Time Frame: Tested 6 to 8 days following patient reporting a positive ovulation test (LH surge). If no surge is detected, progesterone lab will be drawn on Cycle day 21-24.
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate
Number analyzed (Participants) | 98 | 92
Participants | 91 | 89

2. Secondary Outcome: Number of Corpora Lutea
Description: Number of corpora lutea on ultrasound
Time Frame: Cycle day 21-24 of 1st treatment cycle
Population: Participants who completed study ultrasound during c1st study treatment cycle.
Measure: Mean (Standard Deviation); unit: number of corpora lutea
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate
Number analyzed (Participants) | 97 | 91
number of corpora lutea | 0.64 (0.68) | 1.09 (1.02)

3. Secondary Outcome: Number of Corpora Lutea
Description: Number of corpora lutea on ultrasound
Time Frame: Cycle day 21-24 of 2nd treatment cycle
Population: Participants who completed a study ultrasound in their 2nd study treatment cycle.
Measure: Mean (Standard Deviation); unit: number of corpora lutea
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate
Number analyzed (Participants) | 89 | 74
number of corpora lutea | 0.92 (0.70) | 1.07 (0.78)

4. Secondary Outcome: Number of Corpora Lutea
Description: Number of corpora lutea on ultrasound
Time Frame: Cycle day 21-24 of 3rd treatment cycle
Population: Participants who completed a study ultrasound during their 3rd treatment cycle.
Measure: Mean (Standard Deviation); unit: number of corpora lutea
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate
Number analyzed (Participants) | 75 | 64
number of corpora lutea | 0.99 (0.75) | 1.22 (0.90)

5. Secondary Outcome: Endometrial Thickness
Description: Endometrial thickness assessed by ultrasound
Time Frame: Cycle day 21-24 of 1st treatment cycle
Population: Participants completing study ultrasound during their first study treatment cycle
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate
Number analyzed (Participants) | 97 | 91
mm | 8.52 (3.08) | 9.41 (3.10)

6. Secondary Outcome: Endometrial Thickness
Description: Endometrial thickness assessed by ultrasound
Time Frame: Cycle day 21-24 of 2nd treatment cycle
Population: Participants who completed study ultrasound during their 2nd study treatment cycle
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate
Number analyzed (Participants) | 89 | 74
mm | 9.15 (3.09) | 9.32 (2.81)

7. Secondary Outcome: Endometrial Thickness
Description: Endometrial thickness assessed by ultrasound
Time Frame: Cycle day 21-24 of 3rd treatment cycle
Population: Participants who completed study ultrasound during their 3rd study treatment cycle
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate
Number analyzed (Participants) | 75 | 64
mm | 9.11 (3.11) | 9.41 (2.79)

8. Secondary Outcome: Conception
Description: positive serum or urinary test of hCG
Time Frame: 5 weeks after treatment in treatment cycles 1, 2, and 3 (treatment cycle is 24-35 days depending on ovulation)
Reporting Status: Not Posted

9. Secondary Outcome: Clinical Pregnancy
Description: intrauterine pregnancy with fetal heart motion determined by ultrasound
Time Frame: 6 to 7 weeks after treatment in treatment cycles 1, 2, and 3 (treatment cycle is 24-35 days depending on ovulation)
Reporting Status: Not Posted

10. Secondary Outcome: Multiple Gestation
Description: intrauterine pregnancy with more than one fetal heart motion determined by ultrasound
Time Frame: 6 to 7 weeks after treatment in treatment cycles 1, 2, and 3 (treatment cycle is 24-35 days depending on ovulation)
Reporting Status: Not Posted

11. Secondary Outcome: Live Birth
Description: delivery of a live born infant determined by medical record abstraction
Time Frame: 9-10 months following final treatment cycle (treatment cycle is 24-35 days depending on ovulation)
Reporting Status: Not Posted

12. Secondary Outcome: Multiple Birth
Description: delivery of more than one infant determined by medical record abstraction
Time Frame: 9-10 months following final treatment cycle (treatment cycle is 24-35 days depending on ovulation)
Reporting Status: Not Posted

13. Secondary Outcome: Pregnancy Loss
Description: biochemical pregnancy, miscarriage, or ectopic pregnancy determined by ultrasound or medical record abstraction
Time Frame: Through study completion, an average of 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first day of taking study medication through resolution of that treatment cycle, determined by menses, positive pregnancy test, or random start of next cycle. Typically, 3-6 weeks per cycle. Depending on number of cycles completed could range from 3 (single cycle) to 18 weeks (3 cycles).
Description: Participants reported if they had experienced any side effects on daily logs, identifying the side effects they experienced from a list of known medication side effects. They also had the option to enter free text. For each reported side effect, they were asked to rank the severity.
  Serious adverse events included visits to the Emergency room and those which caused marked limitation in activity.
Arm/Group | Letrozole | Letrozole + Clomiphene Citrate
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/92
Serious Adverse Events (participants affected / at risk) | 2/98 | 2/92
Other Adverse Events (participants affected / at risk) | 68/98 | 69/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=98) | Letrozole + Clomiphene Citrate (N=92)
Mood changes (Psychiatric disorders) | 1 | 0
Back pain (General disorders) | 0 | 1
Abdominal pain (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Food borne illness (Gastrointestinal disorders) | 1 | 0 — Nausea, vomiting, diarrhea and fever.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Letrozole (N=98) | Letrozole + Clomiphene Citrate (N=92)
Hot flash (Reproductive system and breast disorders) | 29 | 45
Constipation (Gastrointestinal disorders) | 4 | 15
Headache (Nervous system disorders) | 41 | 47
Abdominal bloating (Reproductive system and breast disorders) | 19 | 25
Nausea (Gastrointestinal disorders) | 31 | 24
Vomiting (Gastrointestinal disorders) | 5 | 6
Upset stomach (Gastrointestinal disorders) | 19 | 21
Mood changes (Psychiatric disorders) | 27 | 29
Visual changes (Eye disorders) | 2 | 2
Fatigue (General disorders) | 30 | 37
Dark Urine (Renal and urinary disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 21
Arthritic pain (Musculoskeletal and connective tissue disorders) | 12 | 9
Dizziness (Nervous system disorders) | 14 | 5
Breast discomfort (Reproductive system and breast disorders) | 13 | 20
Abdominal pain (General disorders) | 28 | 27/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT05206448/Prot_SAP_000.pdf